CLINICAL TRIAL: NCT04150237
Title: Using Simulation to Ensure Basic Competence in Gastroscopy
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Anders Bo Nielsen, Medical Doctor, Odense University Hospital
Other Study IDs: OP_971
Record Dates: First submitted 2019-10-29; First posted 2019-11-04 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Endoscopy; Simulation; Education; Gastroscopy
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Novices: Medical students
  Interventions: Other: Simulation training in gastroscopy
- Intermediates: Endoscopy (EGD) assisting nurses. No prior self-performed endoscopies
  Interventions: Other: Simulation training in gastroscopy
- Experienced: Medical doctors in medical Gastroenterology or surgery, who have self-performed more than 500 EGD
  Interventions: Other: Simulation training in gastroscopy

INTERVENTIONS:
Other: Simulation training in gastroscopy — Simulation-based training with virtual reality simulation at a Simbionix GI-mentor II endoscopy simulator and procedure training on a phantom.

SUMMARY:
The main purpose of this study is to develop and gather validity evidence for a simulation-based test to ensure learning basic competence in gastroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Medical students enrolled at the University of Southern Denmark who have passed their anatomy exam.
* Experienced endoscopy nurses, who have assisted to more than 100 gastroscopies and with no prior self-performed gastroscopies.
* Experienced medical doctors in medical gastroenterology or surgery, who have self-performed more than 500 gastroscopies.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The medical students will be recruited after passing their anatomy exam at the University of Southern Denmark. The endoscopy nurses will be recruited at Odense University Hospital. Medical doctors in medical gastroenterology and surgery will be recruited at the Odense University Hospital, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Simulation gastroscopy test score | 1-hour test
  Test score based on time usage, landmark and pathology recognition

SECONDARY OUTCOMES:
Total time for the diagnostic exercises | 1-hour test
  A total time for two diagnostic virtual reality tests and a test on a phantom
Total time for the tool exercises | 1-hour test
  A total time of virtual reality tests and two tests on a phantom
Total landmark and pathology recognition for the diagnostic exercises | 1-hour test
  Recognition of a total number of 48 landmarks and pathologies

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided